CLINICAL TRIAL: NCT00699348
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous C.E.R.A. for the Maintenance of Haemoglobin Levels in Hemodialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Monthly Intravenous C.E.R.A. (Mircera) in Hemodialysis Participants With Chronic Renal Anemia
Acronym: CARISMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21438; 2007-005799-15 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- C.E.R.A. (Experimental)
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta (C.E.R.A.)

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta (C.E.R.A.) — Intravenous methoxy polyethylene glycol-epoetin beta (C.E.R.A.) at starting dose of 120, 200, or 360 micrograms every 4 weeks for 24 weeks.
  Other Names: Mircera

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of once-monthly administration of intravenous methoxy polyethylene glycolepoetin beta (Mircera) for the maintenance of hemoglobin levels in hemodialysis participants with chronic renal anemia. Participants currently receiving intravenous epoetin alfa or beta or darbepoetin alfa will receive intravenous Mircera at a starting dose of 120, 200 or 360 micrograms/month (based on the erythropoietin stimulating agent [ESA] dose administered on week -1). Subsequent doses will be adjusted to maintain hemoglobin levels within the target range of 10 to12 gram per deciliter (g/dL). The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal anemia;
* Continuous intravenous maintenance erythropoietin stimulating agent (ESA) treatment during previous month;
* Regular long term hemodialysis therapy with the same mode of dialysis for >=3 months.

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months;
* Significant acute or chronic bleeding, such as overt gastrointestinal bleeding;
* Active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Italy (54):
  - Acireale
  - Ancona
  - Anzio
  - Arenzano
  - Ascoli Piceno
  - Avellino
  - Benevento
  - Bollate
  - Borgomanero
  - Brescia
  - Brindisi
  - Cagliari
  - Castellammare di Stabia
  - Catania
  - Cernusco sul Naviglio
  - Chieri
  - Chieti
  - Civitavecchia
  - Cosenza
  - Ferrara
  - Florence
  - Foggia
  - Genova
  - La Spezia
  - Lecco
  - Legnano
  - Lido di Ostia
  - Lodi
  - Lucera
  - Mantova
  - Matera
  - Milan
  - Milazzo
  - Montevarchi
  - Napoli
  - Nocera Inferiore
  - Novara
  - Nuoro
  - Palermo
  - Pavia
  - Perugia
  - Piacenza
  - Pisa
  - Ravenna
  - Reggio Emilia
  - Roma
  - San Daniele del Friuli
  - San Miniato
  - Sassari
  - Taranto
  - Torino
  - Udine
  - Verona
  - Vicenza

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694
- [Derived] Locatelli F, Mandolfo S, Menegato Adorati M, Villa G, Tarchini R, Pizzarelli F, Conte F, Guastoni C, Ricciardi B, Crotta A. Efficacy and safety of once-monthly continuous erythropoietin receptor activator in patients with chronic renal anemia. J Nephrol. 2013 Nov-Dec;26(6):1114-21. doi: 10.5301/jn.5000251. Epub 2013 Sep 13. PMID 24052462

RESULTS

PARTICIPANT FLOW:
Groups:
- C.E.R.A.: Adult participants with chronic renal disease and who had received intravenous epoetin (epoetin alfa, epoetin beta or darbepoetin alfa) maintenance treatment, received (after fulfilling all inclusion/exclusion criteria and 4 weeks stability verification period [Week -4 to Week 0]) intravenous methoxy polyethylene glycolepoetin beta (C.E.R.A.) at starting dose of 120, 200, or 360 microgram (mcg) every 4 weeks for 24 weeks.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 351
Completed | 261
Not Completed | 90
Not completed — Death | 6
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 11
Not completed — Protocol Violation | 10
Not completed — Lack of Efficacy | 8
Not completed — Failure to return | 1
Not completed — Blood transfusion | 24
Not completed — Renal transplantation | 10
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were treated with at least 1 dose of C.E.R.A. and had a safety follow-up, whether withdrawn prematurely or not.
Groups:
- C.E.R.A.: Adult participants with chronic renal disease and who had received intravenous epoetin (epoetin alfa, epoetin beta or darbepoetin alfa) maintenance treatment, received (after fulfilling all inclusion/exclusion criteria and 4 weeks stability verification period) intravenous C.E.R.A. at starting dose of 120, 200, or 360 mcg every 4 weeks for 24 weeks.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 202

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Mean Hemoglobin Concentration Within Plus or Minus (+/-) 1 Gram Per Deciliter (g/dL) of Reference and Within the Target Range
Description: Percentage of participants maintaining the mean hemoglobin concentration within +/- 1.0 g/dL of their reference hemoglobin value and within the target range of 10.0 to 12.0 g/dL during the efficacy evaluation period (EEP) was assessed. The reference hemoglobin value was defined on the basis of the 5 assessments recorded during the stability verification period (SVP) at Weeks -4, -3, -2, -1 and 0. The mean hemoglobin concentration for each individual participant during the EEP (Week 17 to Week 24) was estimated as a time adjusted average.
Time Frame: Week 17 up to Week 24
Population: Per protocol (PP) population included all participants who received at least 1 dose of C.E.R.A. and for whom data for at least 1 follow-up variable was available with the exception of participants who did not fulfill the protocol specified inclusion criteria for this analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 165
percentage of participants | 60.00 [52.10 to 67.54]

2. Secondary Outcome: Change in Hemoglobin Concentration Between Reference SVP and EEP
Description: The mean change of the time adjusted average of hemoglobin from reference value obtained during the SVP (Week -4 up to Week 0) and the value during EEP (Week 17 up to Week 24) was assessed.
Time Frame: Week -4 up to Week 0 and Week 17 up to Week 24
Population: PP Population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 165
g/dL | -0.10 (0.98)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within the Target Range
Description: Percentage of participants maintaining hemoglobin concentration within the target range of 10.0 to 12.0 g/dL during EEP (Week 17 to Week 24) was assessed.
Time Frame: Week 17 up to Week 24
Population: PP population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 165
percentage of participants | 73.94 [66.54 to 80.45]

4. Secondary Outcome: Median Time Spent by Participants With Hemoglobin Concentration in the Target Range During the EEP
Description: Median time spent by participants with hemoglobin concentration within the target range of 10.0 to 12.0 g/dL during the EEP (Week 17 to Week 24) was assessed.
Time Frame: Week 17 up to Week 24
Population: PP population.
Measure: Median (Full Range); unit: days
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 165
days | 44.0 [0.0 to 56.0]

5. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustment
Description: Percentage of participants requiring any adjustment in the dose of study drug during the dose titration period (DTP: Week 1 to Week 16) and EEP (Week 17 to Week 24) was reported.
Time Frame: Week 1 up to Week 16 and Week 17 up to Week 24
Population: PP population.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 165
percentage of participants
  DTP | 70.3
  EEP | 50.9

6. Secondary Outcome: Number of Participants With Red Blood Cell Transfusion During the Study
Description: Number of participant who underwent red blood cell transfusion during the study was reported.
Time Frame: Week -4 up to Week 52
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 351
participants | 38

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: Only adverse events with an onset date after the start of medication were included.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 98/351
Other Adverse Events (participants affected / at risk) | 23/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=351)
Anaemia (Blood and lymphatic system disorders) | 7
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 2
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1
Retinal detachment (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Catheter site haemorrhage (General disorders) | 1
Device malfunction (General disorders) | 1
Pyrexia (General disorders) | 3
Vessel puncture site haemorrhage (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Bronchopneumonia (Infections and infestations) | 2
Campylobacter intestinal infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Oropharyngitis fungal (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 9
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 3
Haemoglobin decreased (Investigations) | 3
Cachexia (Metabolism and nutrition disorders) | 2
Diabetic foot (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Angiopathy (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Necrosis ischaemic (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral ischaemia (Vascular disorders) | 4
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=351)
Hypertension (Vascular disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.